CLINICAL TRIAL: NCT03086980
Title: Automatic Self Transcending Meditation (ASTM) Versus Usual Care in Patients With Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monali Malvankar, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 108387
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma; Depression; Anxiety; Quality of Life
Keywords: health related quality of life; utility; regression
MeSH Terms: conditions — Glaucoma; Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Self Transcending Meditation (Active Comparator): Automatic Self Transcending Meditation is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness.Research suggests that ASTM may help reduce depression and anxiety.
  Interventions: Other: Automatic Self Transcending Meditation
- Treatment as Usual (TAU) (Placebo Comparator): The usual standard of care for patients with glaucoma includes starting them on first line of drugs. Participants will be initiated and maintained on appropriate dosages of such medications as part of standard of care. The usual standard of care also includes an ophthalmic examination measuring best-corrected Snellen VA and pinhole acuities and a follow-up visit once a year.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Automatic Self Transcending Meditation — Automatic Self Transcending Meditation (ASTM) is a class of meditation that helps quiet the mind. Research suggests that ASTM helps reduce depression, anxiety, stress, and may improve health related quality of life. Further, ASTM is easier to learn and to teach.
  Other Names: Sahaj Samadhi Meditation
  Arms: Automatic Self Transcending Meditation
Other: Treatment as Usual — Usual Care will be provided.
  Other Names: Usual Care
  Arms: Treatment as Usual (TAU)

SUMMARY:
Patients with glaucoma will be randomized to Automatic Self Transcending Meditation (ASTM) plus Treatment as Usual (TAU) or TAU alone to assess changes in Health-related quality of life (HRQoL). HRQoL is a vital construct focusing on impact of health on quality of life. HRQoL data is used in economic evaluations, a component of health economics that compares the cost and consequences of alternative courses of action. This helps policy-makers make complex financial decisions. Along with HRQoL we will measure changes in extent of depression as well as anxiety. Previously published data lacks information of HRQoL in patients with glaucoma. Through this study we shall attempt to correlate HRQoL in this population and assess if ASTM confers changes in HRQoL along with depressive and anxiety symptoms.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of irreversible blindness, afflicting an estimated 60.5 million people worldwide. Further, glaucoma is significantly associated with symptoms of depression, altered mood, and anxiety. Meditation, specifically, Automatic Self Transcending Meditation (ASTM) may help reduce depression, anxiety, stress, and may improve quality of life. ASTM is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness. Research suggests that ASTM is easier to learn and to teach. We will offer patients a specific standardized form of ASTM called Sahaj Samadhi Meditation. In this study we shall measure HRQoL of patients with glaucoma in both ASTM and no intervention arms. HRQoL is an essential measure of quality of life related to health; it helps physician identify hidden morbidities in clinical care as well as improves patient-physician communications. However, majority of current ophthalmic literature describes changes in clinical variables with any intervention whilst lacking information on HRQoL. We think there is a high necessity to assess if there is an association between HRQoL and routinely measured clinical data. A primary purpose of this study is to assess if ASTM confers beneficial effects on HRQoL of glaucoma patients compared to a no intervention arm. Additionally, we will assess changes, if any, that ASTM confers on self-reported depression and anxiety symptoms as a secondary outcome measure. PRIMARY HYPOTHESIS: We hypothesize that in patients with glaucoma ASTM + TAU will lead to significant improvement in HRQoL compared to TAU alone from baseline to 24 weeks after the initial ASTM training. SECONDARY HYPOTHESES: We hypothesize that in patients with glaucoma 1) HRQoL is associated with regularly measured clinical variables 2) ASTM+TAU leads to significant improvement in depression and anxiety symptoms at 24 weeks compared to TAU alone 3) The beneficial effects of ASTM on all studied variables will be sustained at 24 weeks post intervention. STUDY DESIGN: We plan to conduct a single-center, single blind longitudinal randomized controlled trial. Research participants will be 142 men and women (71 in each group). STUDY RECRUITMENT: Potential participants with mild to severe glaucoma as well as glaucoma suspects above the age of 18 years will be screened from the office practice of Dr. Hutnik as per inclusion and exclusion criteria by Dr. Hutnik at the Ivey Eye Institute, London, ON. Letter of information (LOI) will be given to potential participants. An ophthalmic examination - offered as a routine care - for each potential participant (i.e., measuring best-corrected Snellen visual acuity (VA) and pinhole acuities) will be conducted. Data on clinical variables such as visual field and optical coherence tomography (OCT) measurements, including central macular thickening, will be obtained. Questionnaire: Patients will undergo a standardized interview performed by a trained interviewer to measure HRQoL using the time trade-off method (TTO). During the first office visit only, also a screening visit, in the interview, patients will be asked demographic questions including age, gender, and associated medical conditions, such as concurrent ocular conditions, ocular disease other than glaucoma, previous ocular surgery, inflammation, intraoperative complications, preoperative ocular pathology, chronic pain, general diseases that could affect the immune system, and actual infection. In addition, patients will be asked about co-morbidities such as, whether they have high blood pressure, diabetes, arthritis, heart condition, stroke, and other non-ocular medical conditions. Further, the following self-rated scales will be administered at the first office visit: Visual Function Questionnaire (VFQ-25), the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), and Community Integration Questionnaire (CIQ). RANDOMIZATION: Participants will be randomized to either ASTM + TAU or TAU alone equally (1:1) using computer generated randomization numbers available at random.org. A telephone number will be available for study concerns/queries. Pre-randomized information will be stored using unique de-identifiers and downloaded on a secure database. It will not be possible to blind participants to intervention status. Outcome assessors and investigators will be blinded to treatment. It will not be possible to blind participants or staff providing treatment to the intervention status. TREATMENT ARMS: 1. ASTM: Following the initial measurements (common to both ASTM and control group), participants in the ASTM group will undergo ASTM training in groups of 10 or more by certified teachers under the supervision of one of the study collaborator at a room in St. Joseph's Hospital or at the Ivey Eye Institute, 268 Grosvenor Street, London, ON. This involves participating in four, 90-120 minute sessions each of four consecutive days. This will be followed by weekly 60-75 minute follow up sessions for 12 weeks and bi-weekly follow-up sessions for 13 to 24 weeks. Participants will be required to attend 75% of weekly, and 80% of bi-weekly sessions. In addition, participants will be asked to practice ASTM at home for 20 minutes twice daily over the study period (24 weeks). Participants will be asked to log practice frequency and any other noteworthy observations in the log sheet provided to them. Further, the following self-rated scales will be administered by a trained rater at the fourth ASTM session (week 0) as well as at weeks 12, and 24: TTO, VFQ-25, PHQ-9, GAD-7. 2. Control Intervention: Participants randomized to control arm (Treatment as Usual, TAU) will continue to receive their treatment as usual including glaucoma medications. They will follow assessment and study procedures as listed below. Following a duration of week 24 into the study participants in TAU arm will also be offered the opportunity to learn ASTM. No study procedures will be applied or any other information collected during this period. STUDY RECRUITMENT: We anticipate to recruit participants at a rate of at least 2 participants/week over a period of 36 weeks allowing attainment of sample size of n=71. There is no obligation for the participants to take part in the study; all participation is voluntary. PRIMARY (HRQoL) measures at first office visit: Patients from both arms will undergo a standardized interview performed by a trained interviewer to measure HRQoL at the first office visit and study visits (week 0, 4, 6, 8, 12, and 24 weeks). SECONDARY OUTCOME MEASURES (first office visit and study visits: week 0, 4, 6, 8, 12, and 24): VFQ-25, PHQ-9, and GAD-7 will be assessed by a trained interviewer at the first office visit plus the study visit days (week 0, 4, 6, 8, 12, and 24). Note that the PHQ-9 and GAD-7 are self-rated scales and participants will be asked to complete these in presence of the rater. ADDITIONAL PROTOCOL CONDITIONS: Individual patients will be withdrawn from the study interventions if it appears that to continue would be deleterious for their mental health or safety. This can be determined by the patient, the treating clinician and/or the research team and will be supported using the PHQ-9 particularly if there is an increase in the score. Variable Specification: A dependent variable is created based on the HRQoL, an interval scale variable taking values between 0.0 and 1.0. Independent variables: Visual acuity in a better-seeing eye, visual field, optical coherence tomography (OCT) measurements, and patients' demographic characteristics, including age, gender, and associated medical conditions are the independent variables. Visual field, optical coherence tomography (OCT) measurements, and patients' demographic characteristics, including age, are considered as continuous variables. Gender is categorized as male and female and associated medical conditions are categorized as "current medical conditions," which includes concurrent ocular conditions, inflammation; "other diseases," which includes ocular diseases other than glaucoma, chronic pain, general diseases that could affect the immune system, and actual infection; and "medical history," which includes previous ocular surgery, preoperative ocular pathology, and intraoperative complications. Data Grouping: Based on BCVA, study participants will be grouped to visual acuity in better seeing eye (group 1, 20/20 to 20/40; group 2, 20/50 to 20/100; group 3, 20/200 to no light perception). Better seeing will be used since a correlation has been shown between utility score and better seeing eye. These 3 groups were chosen since group 1 represents legal driving vision, group 2 represents moderate visual acuity loss, and group 3 represents legal blindness. Data Analysis: As has been done in many other studies, HRQoL will be calculated by dividing the number of years a patient is willing to trade in return for improved quality of life by the estimated numbers of years of remaining life subtracted by 1.0. Mean, standard deviation, and 95% confidence interval for continuous variables such as visual field, OCT measurements, age, and utility value, will be calculated. For categorical variables, visual acuity in the better-seeing eye, gender, and associated medical conditions, proportions will be calculated. The chi-square test statistic for independence will be used to compare unwillingness to trade time in TTO. The unpaired, two-tailed Student t-test will be used to evaluate the effect of visual acuity in the better eye in four groups and gender on mean of time trade-off utility values. Non-response issues: Non-respondent patients' characteristics will be compared with respondent patients,' and if they do not appear to be statistically significantly different, then these results will be generalized to the sample and population. Data will be analyzed using STATA Software (Version 12.0). The unit of analysis is the HRQoL. Univariate and bivariate analysis will be performed for each independent variable against the dependent variable to elicit the impact of each factor on the pattern of HRQoL without adjusting for the effect of other variables. Models will be deemed statistically significant if they are associated with a significant F value (p < 0.01) and if they explain over 15% variability of the dependent variable. Only those independent variables that are statistically significantly associated with the HRQoL (p < 0.05) will be used for model construction. Since the dependent variable is continuous, we plan to use a non-linear regression model to assess the effect of each independent variable on the dependent variable, while controlling for the confounders. Multicollinearity, high correlation between independent variables, and interaction effects will be evaluated for the model. Validation Analysis: Validation will be performed on the developed NLR model. The collected data will be divided into two portions: one portion, called the "main data," will contain 80% of the samples of the total collected utility values and its associated data; the other portion, called the "test data," will contain the remaining 20%. Validation will be done using test data but having the same coefficient values as the main data to calculate the percentage of correct cases.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma suspects or have mild to severe glaucoma
* at least 18 years of age or above
* deemed competent such as no language issues or communication barriers, no self-reported or physician diagnosed mental health disorder besides having depressive and anxiety symptoms
* have sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 30 minutes
* willing and able to attend 4 initial ASTM training sessions and at least 75% of weekly and 80% of bi-weekly follow up sessions
* willing to dedicate 20 minutes twice per day to ASTM practice at their own home.

Exclusion Criteria:

* Actively suicidal as per self-report (scoring 2 or more on item 9 of the PHQ-9) or on assessment by the physician.
* They are currently participating in other similar studies
* Currently practicing any type of formal meditation, mindfulness or breathing techniques regularly
* unable or unwilling to answer survey questions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Health-related quality of life (HRQoL) | First office visit, Week 0, 4, 6, 8, 12, and 24
  HRQoL is an essential measure of quality of life related to health; it helps physician identify hidden morbidity in clinical care as well as improves patient-physician communications. HRQoL will be measured using time trade-off questionnaire.

SECONDARY OUTCOMES:
Visual Function Score | First office visit, Week 0, 4, 6, 8, 12, and 24
  Visual Function score will be measured using Visual Function Questionnaire (VFQ-25).
Depression | First office visit, Week 0, 4, 6, 8, 12, and 24
  Depression is a feeling of severe despondency and dejection. Depression will be measured using the Patient Health Questionnaire (PHQ-9).
Anxiety | First office visit, Week 0, 4, 6, 8, 12, and 24
  Anxiety will be measured using Generalized Anxiety Disorder (GAD-7).

CONTACTS AND LOCATIONS:
Overall Officials: Monali Malvankar, PhD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected in this study will not be available to other researchers (e.g., outside the primary research group). Since the primary research group has the necessary expertise to analyze the data and do not need any outside help.

REFERENCES:
- [Background] Skalicky S, Goldberg I. Depression and quality of life in patients with glaucoma: a cross-sectional analysis using the Geriatric Depression Scale-15, assessment of function related to vision, and the Glaucoma Quality of Life-15. J Glaucoma. 2008 Oct-Nov;17(7):546-51. doi: 10.1097/IJG.0b013e318163bdd1. PMID 18854731
- [Background] Pappa C, Hyphantis T, Pappa S, Aspiotis M, Stefaniotou M, Kitsos G, Psilas K, Mavreas V. Psychiatric manifestations and personality traits associated with compliance with glaucoma treatment. J Psychosom Res. 2006 Nov;61(5):609-17. doi: 10.1016/j.jpsychores.2006.03.050. PMID 17084138
- [Background] Burns JL, Lee RM, Brown LJ. The effect of meditation on self-reported measures of stress, anxiety, depression, and perfectionism in a college population. Journal of College Student Psychotherapy 25(2):132-144, 2011.
- [Background] Schneider RH, Alexander CN, Staggers F, Rainforth M, Salerno JW, Hartz A, Arndt S, Barnes VA, Nidich SI. Long-term effects of stress reduction on mortality in persons > or = 55 years of age with systemic hypertension. Am J Cardiol. 2005 May 1;95(9):1060-4. doi: 10.1016/j.amjcard.2004.12.058. PMID 15842971